CLINICAL TRIAL: NCT02724072
Title: Evaluation of the Thoraflex™ Hybrid Device for Use in the Repair or Replacement of the Ascending Aorta, Aortic Arch and Descending Aorta in an Open Surgical Procedure.
Brief Title: Thoraflex™ Hybrid IDE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bolton Medical (Industry)
Collaborators: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYBRID-002
Record Dates: First submitted 2016-03-18; First posted 2016-03-31 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2020-11

CONDITIONS: Aortic Aneurysm; Aortic Dissection; Aortic Rupture
Keywords: Thoracic Surgery; Aortic Arch; Frozen Elephant Trunk; Performance Goal
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection; Aortic Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thoraflex™ Hybrid Device. (Experimental): Plexus™ 4 and Ante-Flo™ configurations will be included in this study.
  Interventions: Device: Thoraflex™ Hybrid Device

INTERVENTIONS:
Device: Thoraflex™ Hybrid Device — Single-use medical device sterilized by ethylene oxide which is pre-loaded into a delivery system. The device comprises a gelatin sealed vascular graft combined with a stented graft.

SUMMARY:
The study will assess the effectiveness, safety and clinical outcomes of the Thoraflex™ Hybrid Device in the treatment of aortic disease affecting the aortic arch and the descending thoracic aorta, with or without involvement of ascending aorta.

The study will also assess safety and early clinical outcomes in patients who receive an extension procedure within 1 year of Thoraflex™ Hybrid Device implantation.

Lastly the study will assess the safety and clinical outcomes of patients who receive a Thoraflex™ Hybrid Device for treatment of a ruptured aorta.

Patients will be followed for 3 years.

The Primary Endpoint will be freedom from defined Major Adverse Events (MAE) occurring ≤ 1 year post-procedure.

DETAILED DESCRIPTION:
Vascutek Ltd has developed the Thoraflex™ Hybrid Device (Plexus™ 4 and Ante-Flo™) for the open surgical repair or replacement of damaged or diseased vessels of the aortic arch and descending aorta, with or without involvement of the ascending aorta, in cases of aneurysm and/or dissection. The Thoraflex™ Hybrid Device may be considered a development of the Elephant Trunk (ET) grafts with the addition of a stented distal section. In some cases this will allow for a single stage procedure to be carried out, dependent on the length of affected vessel. As the device is fully sealed and has a collar to aid anastomosis, it removes the requirement for in situ sealing and the suturing together of two devices, thereby reducing cardiopulmonary bypass (CPB) time and overall procedure time.

By reducing the procedure time and negating the need for as many subsequent procedures, this method could greatly improve the success of this procedure and may improve patient outcomes.

The ability to treat complex anatomies in addition to reducing procedure and CPB time, justify the investigation of the Thoraflex™ Hybrid Device. Safety and effectiveness data for subjects treated with the Thoraflex™ Hybrid Device will be compared to historical data from subjects treated using standard ET surgical repair.

It is anticipated that up to 83 patients will be recruited over a 14 month period (approximately). Patients will be evaluated at the following time points: Pre-procedure, Implant, Discharge/30 days, 3 months, 12 months, 24 months and 36 months. An additional visit may be performed for patients who undergo an extension procedure within 1 year of Thoraflex™ Hybrid Device implantation.

65 patients will be recruited to the primary study group (maximum 19 per site). An additional group of patients with a ruptured aorta may also be recruited (up to approximately 18 patients across all sites).

A historical control population has been derived from a comparable patient population who received treatment for thoracic aortic disease using the current standard of care, which is the conventional (2-stage) elephant trunk technique. Using data from the comparator population a Performance Goal Target has been set at 57.4%.

The study will be deemed a success if the lower limit of the 95% confidence interval, associated with the proportion of study patients who are free from the defined composite Major Adverse Events (permanent stroke, permanent paraplegia/paraparesis, unanticipated aortic related re-operation and all-cause mortality) at 1 year post procedure, is greater than 57.4%. Only patients included in the main study group will be included in the Performance Goal Analysis; patients recruited into the additional Aortic Rupture group will not be included in the primary endpoint analysis. All patients in the main study group will be included in the analysis regardless of whether or not an extension procedure has been performed.

ELIGIBILITY:
Inclusion Criteria:

Main Study Group (All patients except Aortic Rupture Patients)

* Patient is aged 18 years or over on date of consent
* Patient is willing and able to comply with all study procedures and study visits
* Patient or their legally authorized representative has given written informed consent to participate in study
* Patient satisfies the inclusion criteria for one of the following categories:

A - Patient has acute dissection of the aorta or B - Patient has chronic dissection of the aorta or C - Patient has an aortic aneurysm (including connective tissue disorders)

A. - Patients with acute dissection of the aorta:

•Patient has acute aortic dissection and requires repair or replacement of damaged or diseased vessels of the aortic arch (with or without involvement of the ascending aorta), and the descending aorta requires replacement, or, in the opinion of the investigator, the patient would derive clinical benefit from prophylactic treatment of the descending aorta.

B. - Patients with chronic dissection of the aorta:

•Patient requires repair or replacement of damaged or diseased vessels of the aortic arch and descending aorta with or without involvement of the ascending aorta due to chronic dissection.

And patient satisfies one or more of the following criteria:

* Patient has aortic sinus, or ascending aorta, or aortic arch, or descending aorta diameter ≥5.5cm (including if asymptomatic) or
* Patient has aorta diameter <5.5cm and growth rate ≥0.5cm/year (including if asymptomatic) or
* Patient has ascending aorta diameter ≥4.5cm and requires valve repair or replacement

C. - Patients with an aortic aneurysm (including connective tissue disorders):

•Patient requires repair or replacement of damaged or diseased vessels of the aortic arch and descending aorta with or without involvement of the ascending aorta

And patient satisfies one or more of the following criteria:

* Patient has aortic sinus, or ascending aorta, or aortic arch, or descending aorta diameter ≥5.5cm (including if asymptomatic) or
* Patient has aorta diameter <5.5cm and growth rate ≥0.5cm/year(including if asymptomatic) or
* Patient has ascending aorta diameter ≥4.5cm and requires valve repair or replacement or
* Patient has Marfan syndrome or other genetically mediated disorders with aortic sinus, or ascending aorta, or arch diameter ≥4.5cm, or, the ratio of the maximal ascending or aortic root area (Π r2) in cm2 divided by the patient's height in meters exceeds 10

Inclusion criteria for Patients with Ruptured Aorta only:

* Patient is aged 18 years or over, on date of consent
* Patient or their legally authorized representative is able and willing to give consent to the patient's enrolment in the study
* Patient has either a ruptured thoracic aorta, or, in the experience of the treating surgeon, is at high risk of imminent rupture of the thoracic aorta

Exclusion Criteria:

Main Study Group (All Patients Except Patients with Ruptured Aorta)

* Patient is unfit for open surgical repair involving circulatory arrest
* Patient has known sensitivity to polyester, nitinol or materials of bovine origin
* Patient has a ruptured aorta
* Patient has active endocarditis or an active infective disorder of the aorta
* Patient has an active systemic infection that, in the opinion of the investigator, would compromise the outcome of the surgical procedure
* Patient is enrolled in another active study and has received an investigational product (device, pharmaceutical or biologic) within 6 months prior to the date of the implant or has not reached the primary endpoint of the study
* Patient is female and is pregnant, or planning to become pregnant during the course of the study. Females of childbearing potential must use acceptable methods of contraception.
* Patient has an uncorrectable bleeding anomaly
* Patient has renal failure (defined as dialysis dependent or serum creatinine ≥2.5mg/dL)
* Patient has known sensitivity to radiopaque contrast agents that cannot be adequately pre-treated
* Patient has a co-morbidity causing expected survival to be less than 1 year
* Patient has any other medical, social or psychological problems that in the opinion of the investigator preclude them from receiving this treatment and the procedures and evaluations pre and post procedure

Exclusion criteria for Patients with Ruptured Aorta only:

* Patient has chronic dissection which, in the opinion of the investigator, can be treated electively
* Patient has aneurysmal disease which, in the opinion of the investigator, can be treated electively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are free from composite Major Adverse Events (Permanent stroke, Permanent paraplegia/paraparesis, Unanticipated aortic-related re-operation, All-cause mortality) at 1 year post-procedure | ≤ 1 year post-procedure
  Freedom from the following composite Major Adverse Events (MAE) occurring ≤ 1 year post-procedure:
  * Permanent stroke
  * Permanent paraplegia/paraparesis
  * Unanticipated aortic-related re-operation (excluding re-operation for bleeding)
  * All-cause mortality
  All relevant events will be adjudicated by CEC. Data will be analysed and presented in a binary format (i.e. Freedom from the listed AE's - Yes/No).

SECONDARY OUTCOMES:
Device Technical Success | At exit from OR (i.e. completion of surgical procedure)
  Device Technical Success is defined as:
  * Successful delivery and accurate placement of the intraluminal part of the graft at the intended implantation site and retrieval of the device delivery system, and
  * Patency of the graft (including branches) and absence of device deformations (e.g., kinks) requiring unplanned placement of additional devices within the graft, and
  * No need for unanticipated or emergency surgery (e.g., return to bypass after initial removal of aortic cannula or reversal of heparin) or re-intervention (e.g. placement of additional unplanned endoluminal devices within the frozen segment) related to the device or procedure.
  All of the above criteria are required to be met in order to achieve technical success.
Procedural Success | At discharge/30 days
  Technical Success, with absence of the following:
  * Death
  * Major adverse ischemic events:
    * Paraplegia
    * Paraparesis
    * Disabling stroke
    * New ischemia
    * Distal procedure-related thromboembolic adverse event
  * Aortic and valve complications:
    * Aortic rupture
    * Increase in aortic regurgitation grade of greater than 1
  * General procedure related complications:
    * Peri-procedural myocardial infarction or need for urgent or emergent PCI/CABG
    * New onset renal failure requiring dialysis
    * Renal dysfunction or volume overload requiring ultrafiltration
    * Bowel ischemia requiring surgery or intervention
    * Life-threatening bleed
    * Severe Heart Failure (HF) or hypotension
    * Prolonged Intubation > 48 hours
    * Pseudoaneurysm of any graft surgical suture line
    * Additional unplanned surgical or interventional procedures related to device
  Technical success with absence of all of above criteria is required in order to achieve procedural success.
Treatment Success | At discharge/30 days and all post-procedural intervals
  Device Technical Success, with absence of the following:
  * Aortic enlargement in the region encompassed by the initial lesion
  * Aortic rupture
  * Fistula formation
  * Lesion-related mortality
  * Loss of device integrity
  * Residual or new Type III endoleak
  * The following subset of major adverse events:
    * Disabling stroke within 30 days of the procedure
    * Paraplegia
    * Paraparesis
  Technical success with absence of all of above criteria is required in order to achieve treatment success.
Individual Patient Success | At 1 year
  Treatment Success at one year, and:
  * Post-operative return to normal activities - employment, household activities, social life, and hobbies, and
  * Improved Health Related Quality of Life Measure (HRQoL) - EQ-5D
  Treatment success and the above criteria are required to be met in order to achieve individual patient success.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S Coselli, Principal Investigator — Baylor St. Luke's
Locations (12):
- United States (12):
  - Stanford University Medical Center, Palo Alto, California
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - The Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - NY Presbyterian Weill Cornell, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) Presbyterian, Pittsburgh, Pennsylvania
  - Baylor St. Luke's, Houston, Texas
  - University of Texas Houston- Memorial Hermann Texas Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Thoraflex™ Hybrid device — https://terumoaortic.com/products/hybrid-solutions/